CLINICAL TRIAL: NCT05140720
Title: Assess the Safety and Immunogenicity of Serum Institute of India's PNEUMOSIL® [Pneumococcal Polysaccharide Conjugate Vaccine Adsorbed (10-Valent)] in Healthy Vietnamese Infants and Toddlers, 6 Weeks to 24 Months of Age
Brief Title: Assess the Safety and Immunogenicity of PNEUMOSIL® Vaccine in Healthy Vietnamese Children, 6 Weeks to 24 Months of Age
Acronym: PNEUMOSIL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vabiotech (Industry)
Collaborators: Vietstar Biomedical Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VX.2020.07
Record Dates: First submitted 2021-09-26; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-08

CONDITIONS: Streptococcus Pneumonia; Vaccine Preventable Disease
Keywords: pneumonia; Pneumococcal vaccine; Vaccine; healthy infants and toddlers
MeSH Terms: conditions — Pneumonia; Vaccine-Preventable Diseases

STUDY DESIGN:
Intervention Model Description: This will be an open label, prospective, bridging study. Pneumococcal conjugate vaccine (PCV)-native subjects in three pre-defined age groups will be recruited into the study.
  Age group 1: From 6 weeks - 6 months Age group 2: From 7 months - 11 months Age group 3: From 12 months - 24 months
  Study subjects will be vaccinated with the primary doses. The dose of 0.5 ml of study vaccine has been selected based on the results from previous clinical studies and in compliance with the approval for marketing authorization in India.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 6 weeks - 6 months of age (Experimental): Group 1: Age group from 6 weeks - 6 months
  Interventions: Biological: PNEUMOSIL®
- 7 - 11 months of age (Experimental): Group 2: Age group from 7 - 11 months
  Interventions: Biological: PNEUMOSIL®
- 12 - 24 months of age (Experimental): Group 3: Age group from 12 - 24 months
  Interventions: Biological: PNEUMOSIL®

INTERVENTIONS:
Biological: PNEUMOSIL® — Study subjects will be vaccinated PNEUMOSIL® with the primary doses as described below:
  Group 1: 3 doses, 4 to 8 week interval Group 2: 2 doses, dose interval > 1 month Group 3: 2 doses, dose interval > 2 months

SUMMARY:
The current study provides data necessary to evaluate the safety and immunogenicity of Serum Institute of India's PNEUMOSIL® [Pneumococcal Polysaccharide Conjugate Vaccine Adsorbed (10-Valent)] in Healthy Vietnamese Infants and Toddlers, 6 weeks to 24 months of age. This is an open label, prospective, bridging study.

DETAILED DESCRIPTION:
In this open label, prospective, bridging study, 300 healthy infants and toddlers will be recruited into the study three pre-defined age groups:

Age group 1: From 6 weeks - 6 months Age group 2: From 7 months - 11 months Age group 3: From 12 months - 24 months

Study subjects will be vaccinated PNEUMOSIL® with the primary doses: Age group 1 with 3 doses, Age group 2 and Age group 3 with 2 doses.

Immunogenicity blood sample for Immunoglobulin G (IgG) will be taken in 35 subjects who completed primary dose series.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants or toddlers, based on medical history and clinical assessment, to be without acute or chronic, clinically significant pulmonary, cardiovascular, hepatobiliary, gastrointestinal, renal, neurological, or hematological functional abnormality or illness that requires medical therapy.
2. Infants or toddlers between 6 weeks to 24 months of age at the first dose
3. Voluntary written informed consent by subject's parents to have the subject participate in the study.
4. Subject's parents being able to comprehend and comply with study requirements and procedures and able and willing to complete subject diary, to return with the subject for all scheduled follow-up visits
5. Subjects born full-term with a weight-to-length Z score of ≥ -2 (WHO child growth standard) at enrollment.
6. Subject with an up-to-date minimal vaccination status for age at the time of enrollment as per National Immunization Program.
7. Subject's parents having a readily identifiable place of residence in the study area, being available for the duration of trial participation, with means of telephone contact.

Exclusion Criteria:

1. Use of any investigational medicinal product prior to randomization or planned use of such a product (other than study vaccine) during the period of study participation. Previous vaccination against Streptococcus pneumoniae.
2. History of Streptococcus pneumoniae infection confirmed by culture from a normally sterile site.
3. History of allergic disease or history of a serious reaction to any prior vaccination or known hypersensitivity to any component of the study vaccines. This included such reactions in older siblings and also includes all components of the vaccines of expanded program on immunization.
4. History of anaphylactic shock.
5. Any abnormal (Grade ≥ 1) vital sign. Note: For fever, axillary temperature of ≥ 37.5°C was considered significant and was repeated to determine whether a subject is eligible for randomization. A minimum of 48 hours following resolution of documented fever needed to pass before the subject could be reassessed for eligibility. The last vital sign measurement was used as the baseline value for the study.
6. Any moderate or severe (Grade ≥ 2) acute illness Note: Infants with a Grade 1 acute illness were enrolled at the discretion of the Principal Investigator (PI).

   Note: Subjects with moderate or severe acute illness would return for clinical reassessment; if the illness had sufficiently resolved, they might still qualify for randomization.
7. Chronic administration (defined as more than 14 consecutive days) of immunosuppressant or other immune modifying drugs prior to the administration of the study vaccine, including the use of glucocorticoids. The use of topical and inhaled glucocorticoids will be permitted.
8. History of administration of a non-study pneumococcal vaccine prior to administration of study vaccine or during the course of study participation (other vaccinations of expanded program on Immunization are accepted).
9. Administration of immunoglobulins and/or any blood products or anticipation of such administration during the study period.
10. History of known disturbance of coagulation or blood disorder that could cause anemia or excess bleeding (e.g., coagulation factor deficiencies, severe anemia at birth). Any clearly documented history in a first-degree relative (e.g., parent, sibling) of the same was also exclusionary.
11. History of suspected primary immunodeficiency. Any clearly documented history in a first-degree relative of the same was also exclusionary.
12. Subject had a sibling die of likely sudden infant death syndrome or die suddenly and without apparent other cause or preceding illness in the first year of life.
13. Evidence of a clinically significant congenital abnormality as judged by the PI.
14. History of meningitis, seizures or any neurological disorder.
15. Evidence by history taking alone of exposure to an HIV-positive individual through maternal fetal transmission, breast milk, or other blood-borne mechanisms.
16. Subject being a direct descendant (child or grandchild) of any person employed by the Sponsor, the contract research organization (CRO), the PI, study site personnel, or department.
17. Any medical or social condition that in the opinion of the PI might interfere with the study objectives, pose a risk to the subject, or prevent the subject from completing the study follow-up.

Note: The specific exclusion criteria (e.g., abnormal vital sign, acute illness) were reassessed at all vaccination visits. Any subject who was not vaccinated due to an acute abnormality assessed at the 2nd or 3rd vaccination visit (V2 or V3) would return once the acute issue has resolved. A minimum of 48 hours must have passed after a documented fever before a subject could be vaccinated. This safety requirement was not deemed a protocol deviation if the visit fell outside the vaccination window; however, it was encouraged to maintain the vaccination window whenever possible in these situations.

Ages: 6 Weeks to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2022-01-25 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Percent of participants with immediate solicited adverse events (AEs), serious adverse events (SAEs) at least 30 minutes after each study vaccine administration. | 30 minutes after each vaccination
  The incidence and severity of immediate solicited local and systemic AEs, SAEs at least 30 minutes observation after each dose of the study vaccine.
Percent of participants with solicited AEs, SAEs within 7 days after each study vaccine administration. | within 7 days after each vaccination
  The incidence and severity of solicited local and systemic AEs, SAEs within 7 days after each dose of the study vaccine.
Percent of participants with solicited AEs, SAEs within 28 days after each dose of the study vaccine. | within 28 days after each vaccination
  The incidence and severity of solicited local and systemic AEs, SAEs within 28 days after each dose of the study vaccine
Percent of participants with immediate unsolicited AEs, SAEs at least 30 minutes after each study vaccine administration. | 30 minutes after each vaccination
  The incidence and severity of immediate unsolicited local and systemic AEs, SAEs at least 30 minutes observation after each dose of the study vaccine.
Percent of participants with unsolicited AEs, SAEs until 28 days after the last primary dose. | From the first primary dose to 28 days after the last primary dose vaccination.
  Percent of participants with unsolicited local and systemic AEs, SAEs from the first primary dose to 28 days after the last primary dose vaccination.

SECONDARY OUTCOMES:
Geometric mean (μg/mL) of IgG concentration for each serotype at 28 days after the last primary dose. | at 28 days after the last primary dose.
Proportion of patients achieving seroconversion with IgG > 0.35 μg/mL as defined by WHO at 28 days after the last primary dose. | at 28 days after the last primary dose.

CONTACTS AND LOCATIONS:
Overall Officials: Son T Vu, PhD, Principal Investigator — Vietnam Military Medicine University

IPD SHARING:
Plan to Share IPD: No